CLINICAL TRIAL: NCT02490436
Title: A Randomized, Cross-over, Placebo-controlled, Double-blind, Single-center, Phase II Study of Cetuximab in Patients With Treatment-refractory, Non-malignant Severe Chronic Neuropathic Pain
Brief Title: Novel Treatment Option for Neuropathic Pain
Acronym: NoTOPain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Collaborators: Frontier Science & Technology Research Foundation, Inc. (Industry); Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SFK3 / 062202_281; 2015-001195-21 (EudraCT Number); 2015/618/REK sør-øst D (Other: Regional Committees for Medical and Health Research Ethics)
Record Dates: First submitted 2015-06-05; First posted 2015-07-03 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Neuralgia; Complex Regional Pain Syndromes
MeSH Terms: conditions — Neuralgia; Complex Regional Pain Syndromes | interventions — Cetuximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: active drug first (Experimental): Cetuximab in treatment period 1, placebo in treatment period 2, and open-label cetuximab in treatment period 3.
  Interventions: Drug: Cetuximab; Drug: Placebo
- B: placebo first (Experimental): Placebo in treatment period 1, cetuximab in treatment period 2, and open-label cetuximab in treatment period 3.
  Interventions: Drug: Cetuximab; Drug: Placebo

INTERVENTIONS:
Drug: Cetuximab — Randomized cross-over between cetuximab and placebo
  Other Names: Erbitux
Drug: Placebo — Randomized cross-over between cetuximab and placebo

SUMMARY:
The purpose of this study is to determine whether the EGFR-inhibitor cetuximab is better than placebo for the treatment of neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent and anticipated compliance.
* Pain defined as "definite" neuropathic pain, according to the Special Interest Group on Neuropathic Pain guidelines or defined as "probable" NP, according to the guidelines, if the confirmatory test was a positive diagnostic test. Complex regional pain syndrome can be included despite lack of an offending lesion, as long as the "Budapest criteria" are fulfilled
* Neuropathic Pain associated with compressive nerve states (including failed surgery) or CRPS (according to the "Budapest criteria")
* PainDETECT score of at least 13 with average pain intensity of at least 6 /10 over the last four weeks. In addition, a painDETECT pattern indicating that the underlying neuropathic pain is constantly present.
* Worst pain intensity higher than 6 for five of seven days during the screening phase, according to Brif Pain Inventory.
* The patient should be able to distinguish between the neuropathic pain and other pain conditions, including elements of nociceptive pain caused by the same disease process.
* Neuropathic pain duration of between six and thirty months, deemed chronic and likely to be irreversible by clinical history and findings.
* No new or increased neuropathic pain treatment for the last four weeks.
* Standard medical treatments for the patients' underlying condition or neuropathic pain must have been considered or tried and must, according to the opinion of the referring or a consulted pain specialist, be judged to be inappropriate or of insufficient potential efficacy.
* Referring physician agreement to follow up the patient after study completion according to the best possible and available pain treatment and care.
* Women of childbearing potential and men must use an acceptable method of contraception throughout the study, and for 30 days after the last study drug administration.
* Negative pregnancy test within 7 days before each treatment period where appropriate.
* White blood cell count ≥ 3 × 109 with neutrophils ≥ 1.5 × 109/L, platelet count ≥ 100 × 109/L and hemoglobin ≥ 6.21 mmol/L (10 g/dL). Total bilirubin ≤ 1.5 × upper limit of reference range and AST and ALT ≤ 2.5 × upper limit of reference range within the last 28 days before inclusion.
* Aged 18 or above

Exclusion Criteria:

* Neuropathic pain origin in the central nervous system.
* Phantom limb pain or a significant component of nociceptive pain.
* Ascending distal small fiber peripheral neuropathy.
* Patients primarily experiencing pain 'attacks', i.e. pattern of neuropathic pain depicted in picture 3 of the painDETECT.
* Other pain state that may interfere with evaluation of the studied neuropathic pain condition.
* Any underlying medical or psychiatric condition, clinical disorder or laboratory finding, which in the opinion of the investigator may interfere with study objectives.
* Uncontrolled or unstable diabetes.
* Severe or uncontrolled cardiovascular disease (congestive heart failure NYHA III or IV), unstable angina pectoris, history of myocardial infarction within the last twelve months, significant arrhythmias
* Severe cerebrovascular disease during the six months prior to inclusion.
* Active and ongoing eye and skin disorders or newly diagnosed gastric ulcer that may interfere with the study treatment.
* History of allergic reaction to any of the study treatment components, red meat or tick bites.
* Previous treatment with any EGFR-pathway inhibitor.
* Women who are pregnant or breastfeeding.
* Participation in another clinical trial within the past 90 days.
* Use of any investigational agent within 90 days prior to day 1 of study drug.
* Known drug abuse/alcohol abuse, legal incapacity or limited legal capacity or any other reason that, in the opinion of the investigator precludes the subject from participating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change in average neuropathic pain score using an 11-point numeric rating scale. | Days 4-8 after each infusion of cetuximab and placebo

SECONDARY OUTCOMES:
Comparison of frequency, in all patients on active treatment of at least a 30% reduction of average neuropathic pain score using an 11-point numeric rating scale. | Days 4-8 after each infusion of cetuximab and placebo
Comparison of frequency in all patients on active treatment of at least a 50% reduction of average neuropathic pain score using an 11-point numeric rating scale. | Days 4-8 after each infusion of cetuximab and placebo
Comparison of change in average worst neuropathic pain score using an 11-point numeric rating scale. | Days 4-8 after each infusion of cetuximab and placebo
Comparison of frequency, in all patients on active treatment of at least a 30% reduction of average worst neuropathic pain score using an 11-point numeric rating scale. | Days 4-8 after each infusion of cetuximab and placebo
Comparison of frequency in all patients on active treatment of at least a 50% reduction of average worst neuropathic pain score using an 11-point numeric rating scale. | Days 4-8 after each infusion of cetuximab and placebo
Patient Global Impression of Change. | 7 days after each infusion.
Brief Pain Iinventory (short form) interference scores, comparing cetuximab to the placebo. | Days 4-8 after each infusion during treatment periods 1 and 2.
Brief Pain Iinventory (short form) total scores, comparing cetuximab to the placebo. | Days 4-8 after each infusion during treatment periods 1 and 2.
2-hourly waking time 11-point numeric rating scale (item #6 from the Brief Pain Inventory) in the first 24 hours and daily thereafter. | 2-hourly in first 24 hours after infusion and daily thereafter until end of study (day 86).
Number of AE and SAE recording | From signing informed consent (within 28 days prior to first study treatment) and until 30 days after the last study infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Kersten, MD PhD, Principal Investigator — Center for Cancer Treatment, Sørlandet Hospital, Kristiansand
Locations (1):
- Center for Cancer Treatment, Sorlandet Hospital HF, Kristiansand, Norway

REFERENCES:
- [Derived] Kersten C, Cameron MG, Bailey AG, Fallon MT, Laird BJ, Paterson V, Mitchell R, Fleetwood-Walker SM, Daly F, Mjaland S. Relief of Neuropathic Pain Through Epidermal Growth Factor Receptor Inhibition: A Randomized Proof-of-Concept Trial. Pain Med. 2019 Dec 1;20(12):2495-2505. doi: 10.1093/pm/pnz101. PMID 31106835